CLINICAL TRIAL: NCT03524430
Title: RNA Disruption Assay (RDA)-Breast Cancer Response Evaluation for Individualized Therapy (BREVITY / BREVITY-02 in Germany)
Brief Title: RNA Disruption Assay (RDA)-Breast Cancer Response Evaluation for Individualized Therapy
Acronym: BREVITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rna Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RnaDx-BRV-BC- 01; RnaDx-BRV-BC- 02 (for Germany) (Other: Rna Diagnostics Inc.)
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasm Female
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Masking Description: This is a diagnostic study. The RDI operator that assesses patient response to therapy using the RDA test is blinded to patient outcome. The clinicians and patients will not receive the RDI score in order to not act on the RDA test result (because this is an investigational study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Interventional Study Arm (Experimental): There will be 2 biopsy collection time points with 2 core needle biopsy specimens taken at each biopsy collection time point for RDA analysis during neoadjuvant chemotherapy.
  Interventions: Procedure: Core needle biopsy

INTERVENTIONS:
Procedure: Core needle biopsy — 1st core needle biopsy for RDA (2 specimens): Time Point: 35 +/-4 days after initiation of chemotherapy.
  If no change is made to the therapy, a second biopsy (2 specimens) will be performed at 55 +/- 5 days after therapy initiation.
  If there is a change of drugs, the second biopsy (2 specimens) will be performed at ~2-3 weeks after initiation of new drugs; Timing by type of drug schedule 3-weekly: at 16 days +/- 2 days, Bi-weekly: at day of 2nd dose preferably before drug admin., Weekly: at day of 4th dose preferably before drug admin.

SUMMARY:
The current study aims to provide validation results of RNA Disruption Assay (RDA) as a tumour response assessment tool that uses tumour core biopsies taken starting from 35 +/- 4 days after the initiation of neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Study Rationale:

There is some evidence that identifying non-responders early in neoadjuvant treatment and offering alternative agents (response-guided therapy) increased pathological complete response (pCR) rates and/or survival resulting in improved care and incremental cost effectiveness.

Differentiating non-responders to chemotherapy from responders with reliable guidance tools early during therapy is crucial to the success of response-guided therapy.

The current study aims to provide validation results of RDA as a tumor response assessment tool that uses tumor core biopsies starting from 35 +/- 4 days after the initiation of neoadjuvant chemotherapy.

Study Objectives and Endpoints:

The primary objective of the study is to determine the 2 RDI cut-offs to have a diagnostic test optimized in terms of both negative and positive predictive values NPV and PPV (in a training set of patients i.e. phase 1 of the study) for predicting nopCR/pCR and to establish the performance characteristics for the first cut-off (test result "zone 1") in terms of NPV as primary endpoint (in a validation set i.e. phase 2).

The secondary objective is to assess the test's NPV in the different cancer subtypes and the test's PPV in Her2+ patients; also to assess and compare pCR prevalence, residual cancer burden (RCB class at surgery) and DFS (secondary endpoints) in zones 1-3 for all patients and each cancer subtype.

Patient Population:

The study aims to enroll approximately 801 patients in centers in the US, Canada, Italy, Germany, Spain and France and Poland.

The population consists of patients diagnosed with invasive breast cancer and scheduled to receive neoadjuvant chemotherapy as part of standard of care treatment. Throughout the study, patients will receive standard of care neoadjuvant chemotherapy treatments including taxanes, anthracyclines or other targeted drugs and drug combinations as prescribed based on the investigators' / clinicians' choice. Adjuvant therapies (e.g. radiotherapy, hormonal treatment … etc.) may be prescribed to patients according to standard of care and independently of the RDI score results.

RDA is presently in an experimental stage and clinicians will not receive or use the RDA results in this study.

Biopsy Collection:

* 1st core needle biopsy for RDA (2 specimens): Time Point: 35 +/- days after initiation of neoadjuvant chemotherapy;
* 2nd core needle biopsy for RDA (2 specimens): Time Point: if therapy is changed (as part of SoC), a second biopsy ~2-3 weeks after initiation of new drugs; Timing by type of drug schedule 3-weekly: at 16 days +/- 2 days, Bi-weekly: at day of 2nd dose preferably before drug admin., Weekly: at day of 4th dose preferably before drug admin. If Therapy is not changed (as part of SoC), a second biopsy is taken at 55 +/- 5 days after the first initiation of neoadjuvant therapy.

Statistical Plan:

The study consists of a training set / phase 1 (80 fully evaluable patients) to determine response zone cut-offs using pCR outcomes and RDA's predictive values, and a validation set / phase 2 (454 fully evaluable patients) to validate the performance characteristics of the RDA test. The study aims to enroll 801 patients in order to achieve an accrual of 534 fully evaluable patients (phase 1 and 2) which is the number required to adequately statistically power the trial. Recruitment per subgroup of cancer subtypes will be closed when the target number of fully evaluable patients per subgroup is reached for both phase 1 and 2. Combined statistical analysis and various subgroup analyses will be performed for the primary and secondary objectives.

Duration and Follow-up:

There will be an active patient accrual until last patient is accrued (to achieve the required fully evaluable patient numbers) in addition to 60 months of patient follow-up.

ELIGIBILITY:
Inclusion Criteria

* Women aged at least 18 years;
* Patients must be able to provide informed consent and sign the informed consent form to participate in the RDA study before any study procedures starts;
* Newly diagnosed clinical stage I, II or III breast cancer with complete surgical excision of the breast cancer after neoadjuvant therapy as the treatment goal;
* Tumour size at least 1 cm in one dimension by clinical or radiographic exam (WHO criteria);
* Must have histological confirmation of invasive breast cancer of any subtype or grade;
* Patient is scheduled for neoadjuvant chemotherapy +/- antibodies and +/- other drugs according to Standard of Care;
* Patient willing to have 2 research core needle biopsies (for RDA) taken at 2 collection timepoints during neoadjuvant chemotherapy treatment.

Exclusion Criteria

* Patient who has had prior local (i.e. surgery or radiotherapy) or systemic (i.e. endocrine or cytotoxic) therapy for the current breast cancer;
* Participation in another interventional clinical trial with concurrent treatment with experimental drugs to treat the current breast cancer during the period of neoadjuvant therapy (from diagnosis until surgery);
* Stage IV breast cancer;
* Bilateral or multicentric breast tumour;
* Prior malignant disease except curatively treated in-situ maligancies;
* Concurrent pregnancy;
* Breast feeding woman;
* Concurrent medical, psychiatric or addictive disorders that may limit the ability to give informed consent or complete the trial;
* Reasons indicating risk of poor compliance with study procedures;
* Patient not able to consent;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | At surgery after completion of neoadjuvant therapy
  (ypT0,ypN0) / (ypTis,ypN0)

SECONDARY OUTCOMES:
Disease-free survival | 5 years of survival follow-up
  Time between diagnosis and first event of progression or death
Residual Cancer Burden | At surgery
  RCB Class

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Trudeau, MD, Principal Investigator — Sunnybrook Health Sciences Center, Toronto, Canada; Daniele Generali, MD, Principal Investigator — SST di Cremona Multidisciplinare di Patologia Mammaria, Italy; Foluso Ademuyiwa, MD, Principal Investigator — Washington University School of Medicine, St Louis, USA; Thierry Petit, MD, Principal Investigator — Institut de Cancérologie, Strasbourg, France; Joke Tio, MD, Principal Investigator — Munster, Germany; Eva Ciruelos, MD, Principal Investigator — Madrid, Spain; Tomasz Jankowski, MD, Principal Investigator — NZOZ Neuromed, Lublin, Poland
Locations (7):
- Siteman Cancer Center, St Louis, Missouri, United States
- Sunnybrook Health Sciences Center, Toronto, Canada
- Institut de Cancerologie de Strasbourg, Strasbourg, France
- Universitätsklinikum Münster, Münster, Germany
- SST di Cremona Multidisciplinare di Patologia Mammaria, Italy, Cremona, Italy
- NZOZ Neuromed, Lublin, Poland
- Hospital U. 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parissenti AM, Guo B, Pritzker LB, Pritzker KP, Wang X, Zhu M, Shepherd LE, Trudeau ME. Tumor RNA disruption predicts survival benefit from breast cancer chemotherapy. Breast Cancer Res Treat. 2015 Aug;153(1):135-44. doi: 10.1007/s10549-015-3498-9. Epub 2015 Jul 25. PMID 26208483
- [Background] Narendrula R, Mispel-Beyer K, Guo B, Parissenti AM, Pritzker LB, Pritzker K, Masilamani T, Wang X, Lanner C. RNA disruption is associated with response to multiple classes of chemotherapy drugs in tumor cell lines. BMC Cancer. 2016 Feb 24;16:146. doi: 10.1186/s12885-016-2197-1. PMID 26911141
- [Background] Toomey S, Eustace AJ, Pritzker LB, Pritzker KP, Fay J, O'Grady A, Cummins R, Grogan L, Kennedy J, O'Connor D, Young L, Kay EW, O'Donovan N, Gallagher WM, Kalachand R, Crown J, Hennessy BT. RE: RNA Disruption Assay as a Biomarker of Pathological Complete Response in Neoadjuvant Trastuzumab-Treated Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer. J Natl Cancer Inst. 2016 Jul 4;108(8):djw111. doi: 10.1093/jnci/djw111. Print 2016 Aug. No abstract available. PMID 27377904
- [Background] Pritzker K, Pritzker L, Generali D, Bottini A, Cappelletti MR, Guo B, Parissenti A, Trudeau M. RNA Disruption and Drug Response in Breast Cancer Primary Systemic Therapy. J Natl Cancer Inst Monogr. 2015 May;2015(51):76-80. doi: 10.1093/jncimonographs/lgv015. PMID 26063893
- [Result] Cazzaniga ME, Ademuyiwa F, Petit T, Tio J, Generali D, Ciruelos EM, Califaretti N, Poirier B, Ardizzoia A, Hoenig A, Lex B, Mouret-Reynier MA, Giesecke D, Isambert N, Masetti R, Pitre L, Wrobel D, Augereau P, Milani M, Rask S, Solbach C, Pritzker L, Noubir S, Parissenti A, Trudeau ME. Low RNA disruption during neoadjuvant chemotherapy predicts pathologic complete response absence in patients with breast cancer. JNCI Cancer Spectr. 2024 Jan 4;8(1):pkad107. doi: 10.1093/jncics/pkad107. PMID 38113421